CLINICAL TRIAL: NCT01789892
Title: FDG PET/CT: Reducing False Positive Mediastinal Uptake by Premedicating With Methylprednisolone
Brief Title: Methylprednisolone Before Fludeoxyglucose-Labeled Positron Emission Tomography in Patients With Lung Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no patient accrual
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: OSU-10012; NCI-2012-00530 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Methylprednisolone; Methylprednisolone Acetate; Methylprednisolone Hemisuccinate; Fluorodeoxyglucose F18; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (methylprednisolone and FDG PET/CT scan) (Experimental): Within 1-14 days of undergoing standard FDG PET/CT scan, patients receive methylprednisolone IV and then undergo a second FDG PET/CT scan.
  Interventions: Drug: methylprednisolone; Radiation: fludeoxyglucose F 18; Procedure: positron emission tomography; Procedure: computed tomography

INTERVENTIONS:
Drug: methylprednisolone — Given IV
  Other Names: Depo-Medrol; Medrol; MePRDL; Solu-Medrol; Wyacort
Radiation: fludeoxyglucose F 18 — Undergo FDG PET/CT scan
  Other Names: 18FDG; FDG
Procedure: positron emission tomography — Undergo FDG PET/CT scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo FDG PET/CT scan
  Other Names: tomography, computed

SUMMARY:
The purpose of this study is to determine whether giving an anti-inflammatory medication (corticosteroid) prior to a positron emission tomography scan (PET) scan may reduce or eliminate false findings related to inflammation

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess whether premedication with a corticosteroid may reduce false positive findings on fluorodeoxyglucose (fludeoxyglucose F 18 [FDG[) PET/computed tomography (CT) scans in lung cancer patients, by reducing radiotracer uptake in thoracic lymph nodes related to inflammation.

OUTLINE:

Within 1-14 days of undergoing standard FDG PET/CT scan, patients receive methylprednisolone intravenously (IV) and then undergo a second FDG PET/CT scan.

After completion of study treatment, patients are followed up for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing initial staging of biopsy proven lung cancer (all cancer stages included)
* Undergone clinical FDG PET/CT scan within 14 days of enrollment

Exclusion Criteria:

* Prisoners
* Diabetic patients (on insulin, on oral hypoglycemic, or fasting glucose > 180 mg/dl)
* Serious infection within 14 days of enrollment
* Known hypersensitivity to methylprednisolone
* Viral skin lesions
* Immunocompromised ANC(absolute neutrophil count < 1000/microliter)
* Pregnant/nursing
* History of tuberculosis or systemic fungal disease
* History of steroid psychosis
* Current peptic ulcer disease or diverticulitis
* Corticosteroid use within 14 days of enrollment (including inhaled steroids)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Continuous standardized uptake values (SUV) | Within 1-14 days of first scan
  The SUV on the first and second PET scans will be recorded and summarized on a receiver operating characteristic (ROC) curve. We will explore the ROC curve for percent change in SUV or uptake ratio from the first to the second scan. We will explore thresholds for SUV and uptake values on the ROC curve by determining the values of acceptable combinations of true positive fractions (TPF) and false positive fractions (FPFs). We will use regression methods to adjust for possible confounding patient demographics, disease severity and disease history.

CONTACTS AND LOCATIONS:
Overall Officials: David Barker, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu